CLINICAL TRIAL: NCT04911374
Title: An Open-Label Clinical Study to Evaluate the Efficacy and Tolerability of a Multi-Ingredient Anti-aging Face Moisturizer and Eye Cream Targeting Aging
Brief Title: An Open-Label Clinical Study to Evaluate the Efficacy of a Face Cream and Eye Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C20-D134
Record Dates: First submitted 2021-05-21; First posted 2021-06-03 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Wrinkle; Photoaging; Fine Lines

STUDY DESIGN:
Intervention Model Description: Open-label study. 45 female subjects recruited, 35 to 65 years, Fitzpatrick skin type I-VI, with mild to moderate droopy eyelids, moderate crow's feet wrinkles, and moderate global photodamage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-Aging Face Moisturizer and Eye Cream (Other): Dual Regimen:
  1. Multi-ingredient anti-aging face moisturizer
  2. Multi-ingredient anti-aging eye cream
  Interventions: Other: Gentle Cleansing Lotion, Revision Skincare; Other: Aveeno Face Milk SPF 40+

INTERVENTIONS:
Other: Gentle Cleansing Lotion, Revision Skincare — Gentle cleansing lotion to be used by study participants
Other: Aveeno Face Milk SPF 40+ — Sunscreen to be applied after application of face moisturizer and eye cream in the morning. Participants were asked to apply the sunscreen if sun exposure was more than 30 minutes per day.

SUMMARY:
This single-center clinical trial is being conducted to assess the efficacy and tolerability of an anti-aging eye cream and face moisturizer when used over the course of 12 weeks twice-daily by women, 35-65 years, with mild to moderate droopy eyelids, moderate crow's feet wrinkles, and moderate global facial photodamage.

DETAILED DESCRIPTION:
This was an institutional review board (IRB)-approved study. Female subjects, 35-65 years of age, Fitzpatrick skin type I-VI, with mild to moderate droopy eyelids, moderate crow's feet wrinkles, and moderate global photodamage were recruited. Subjects applied a multi-ingredient anti-aging face moisturizer and eye twice-daily for 12 weeks. Subjects were provided with a gentle cleansing lotion and a sunscreen SPF 40+ to be utilized during the course of the study.

Clinical grading of efficacy and tolerability parameters, VISIA-CR imaging, raking light VISIA analysis, skin pH, Tewameter, and pinch recoil measurements were performed at baseline, weeks 4, 8, and 12. Optical coherence tomography (OCT) imaging was performed at baseline and week 12.

A total of 42 subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35 and 65 years
* Women with Fitzpatrick skin type I-VI
* Subjects must have mild to droopy eyelids, moderate crow's feet wrinkles, and moderate photodamage
* Subjects must have no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Subjects must be willing to provide verbal understanding and written informed consent.

Exclusion Criteria:

* Subjects which had a health condition and/or pre-existent dormant dermatological disease on the face
* Subjects that had any invasive or non-invasive skin treatments, or invasive medical procedures three months prior to the study
* Subjects that are unwilling to comply with the protocol
* Female subjects who are pregnant, breast feeding, or planning a pregnancy.
* Subjects who have any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin, including rosacea, acne, and excessively oily or dry skin.
* Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
* Subjects use of any medications that are known to potentially cause changes in the facial skin as determined by the Investigator.
* Subjects who spend excessive time out in the sun.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Improvement of Clinical Efficacy Parameters at 4, 8, and 12 weeks versus Baseline | 12 weeks
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale. A change in scores at week 4, week 8 and week 12 in comparison to baseline indicates an improvement for the indicated parameter.
  The efficacy parameters will be assessed globally on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition): 0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9 = severe (worst possible condition). The lower the score equates to the best possible outcome.
Lack of Significant Increase in Objective Tolerability Parameters at week 4, 8, 12 compared to Baseline | 12 weeks
  The primary tolerability endpoint will be the Investigator Tolerability Assessment of Erythema, Edema and Dryness. A change in scores or lack of significant change at week 4, week 8 and week 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example for Erythema: Erythema 0 = None No erythema of the treatment area
  1. = Mild Slight, but definite redness of the treatment area
  2. = Moderate Definite redness of the treatment area
  3. = Severe Marked redness of the treatment area

SECONDARY OUTCOMES:
Lack of Significant Increase in Subjective Tolerability Parameters at week 4, 8, 12 compared to Baseline | 12 weeks
  The secondary tolerability endpoint will be the Subject Tolerability Assessment of Burning, Itching and Stinging. A change in scores or lack of significant change at week 4, week 8 and week 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example Burning. 0 = None No burning of the treatment area
  1. = Mild Slight burning sensation of the treatment area; not really bothersome
  2. = Moderate Definite warm, burning of the treatment area that is somewhat bothersome.
  3. = Severe Hot burning sensation of the treatment area that causes definite discomfort and may interrupt daily activities and/or sleep
Decrease in transepidermal water loss at weeks 4, 8, and 12 versus baseline | 12 weeks
  • Tewameter Measurements at baseline and weeks 4, 8, and 12. A change in Tewameter values reflects an improvement in the barrier properties of the skin; an absence of a change in treated skin indicates mildness of the applied treatment.
Stable skin pH during 12 week study | 12 weeks
  •pH Measurements at baseline and weeks 4, 8, and 12. A stable pH measurement reflects that the test product does not affect the overall cutaneous pH value.
Improvement in Epidermal Thickness after 12 weeks versus baseline | 12 weeks
  •OCT Imaging Procedures at baseline and week 12, with image analysis performed at the end of the study using images from baseline and week 12. A change in epidermal thickness indicates improvement.

OTHER OUTCOMES:
Self-Assessment Questionnaire | 12 weeks
  The secondary efficacy endpoints will be the Self-Assessment Questionnaire and the Subject Treatment Satisfaction and Ease of Use Questionnaire. A change in response values at week 4, week 8 and week 12 indicates an improvement compared to baseline response values. Subjects are asked to rate based on a scoring system of the following: from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement/ question being asked.

CONTACTS AND LOCATIONS:
Locations (1):
- Stephens and Associates, Richardson, Texas, United States